CLINICAL TRIAL: NCT03838081
Title: Evaluation the Effect of Verbal & Written Information and the Previous Surgical Experience on the Anxiety of Third Molar Extraction
Brief Title: Evaluation on the Anxiety of Third Molar Extraction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Kevser Sancak, Oral and Maxillofacial surgery, Principal investigator, Ankara University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 36290600/69
Record Dates: First submitted 2019-02-10; First posted 2019-02-12 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Dental Anxiety
Keywords: third molar extraction; Preoperative anxiety; Dental Anxiety

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): Group 1: Patients who were given only basic information verbally
  Interventions: Behavioral: Spielberger State Anxiety Inventory (STAI-S),; Behavioral: Dental Fear Scale (DFS); Behavioral: Modified Dental Anxiety Scale (MDAS); Behavioral: Visual Analog Scale (VAS)
- Group 2 (Experimental): Group 2: Patients with detailed written information about preoperative, intraoperative, and postoperative periods
  Interventions: Behavioral: Spielberger State Anxiety Inventory (STAI-S),; Behavioral: Dental Fear Scale (DFS); Behavioral: Modified Dental Anxiety Scale (MDAS); Behavioral: Visual Analog Scale (VAS)
- Group 3 (Experimental): Group 3: Patients with previous experience and knowledge about third molar extraction
  Interventions: Behavioral: Spielberger State Anxiety Inventory (STAI-S),; Behavioral: Dental Fear Scale (DFS); Behavioral: Modified Dental Anxiety Scale (MDAS); Behavioral: Visual Analog Scale (VAS)

INTERVENTIONS:
Behavioral: Spielberger State Anxiety Inventory (STAI-S), — STAI is one of the most frequently used scales in anxiety research, although it is not a specific scale for dental anxiety
Behavioral: Dental Fear Scale (DFS) — DFS is a scale developed by Kleinknecht used to determine dental fear in different dimensions. This is a Likert-type scale with a score of 1-5. It has 20 items. It examines the level of fear in terms of dentist avoidance, somatic symptoms of fear, and fear of various applications in dentistry practice
Behavioral: Modified Dental Anxiety Scale (MDAS) — MDAS was developed by Humphris et al. by adding a question related to injection. The scale consists of five-point Likert-type rating with five options. The scoring in this scale varies between 5 and 25
Behavioral: Visual Analog Scale (VAS) — VAS is ideal for evaluating situations that cannot be measured using digital and oral information. In the present study, a scale comprising 100-mm closed-end line was used to measure the anxiety level. One end of the scale was labeled as "no anxiety" and the other end as "maximum anxiety imaginable

SUMMARY:
This study was performed on 66 patients who were admitted for third molar extraction under local anesthesia. The patients were divided into three groups: group 1 with verbal information, group 2 with written information, and group 3 with previous surgical experience. Spielberger State Anxiety Inventory (STAI-S), Dental Fear Scale (DFS), Modified Dental Anxiety Scale (MDAS), and Visual Analog Scale (VAS) were used pre- and postoperatively to evaluate dental anxiety

DETAILED DESCRIPTION:
This prospective study included 66 patients who underwent third molar extraction under local anesthesia in the Oral and Maxillofacial Department, Faculty of Dentistry, Ankara University, Turkey, between September and November 2018. The research protocol was approved by the ethical committee of the institute (No: 36290600/69), Ankara University, Turkey.

Spielberger State Anxiety Inventory (STAI-S), Dental Fear Scale (DFS), Modified Dental Anxiety Scale (MDAS), and Visual Analog Scale (VAS) are commonly used questionnaires for dental anxiety. The latter asked only about age and sex. They were used together before and immediately after surgery to obtain better results in this study.

After examining the panoramic radiographs, patients who underwent extraction were included in Classes 1 and II, Positions A and B according to Pell-Gregory 16 classification, and mesioangular and vertical positions according to the Winter 17 classification.

Each patient was examined by the researcher. The patients were informed about the procedure, and written informed consent was obtained from the patient's preoperative assessment clinic. If a patient had additional questions, they were included as part of the investigation.

The patients were divided into three groups:

Group 1: Patients who were given only basic information verbally Group 2: Patients with detailed written information about preoperative, intraoperative, and postoperative periods Group 3: Patients with previous experience and knowledge about third molar extraction Previous experience was determined before giving the questionnaires. The patients were randomly assigned to group 1 or 2 using an online random allocation software (www.randomization.com). Information was provided on how to complete questionnaires. STAI-S, MDAS, DFS, and VAS were applied to all patients 15 min before the surgery in the waiting room. The demographic data section (age and sex) in the form was filled out by the researcher.

The surgery was carried out under local anesthesia, with no pharmaceutical premedication or sedation. The surgical procedures were performed by a single experienced surgeon in the oral surgery clinic. After the surgery was completed, the patients were taken to the waiting room, and prescribed medications were given. STAI-S, MDAS, DFS, and VAS were reapplied after the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-80 years
* American Society of Anesthesiologists physical status score I and II
* Patients without any systemic disease, or regular medication use.

Exclusion Criteria:

* İnability to read and understand Turkish
* Significantly impaired eyesight or hearing, an existing psychiatric disorder
* Patients aged less than 18 years

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2018-09-15 (Actual); Primary Completion 2018-12-15 (Actual); Study Completion 2019-01-05 (Actual)

PRIMARY OUTCOMES:
Evaluation of anxiety with Spielberger State Anxiety Inventory(STAI-S) between groups preoperatively and postoperatively | 2 minutes
  Spielberger State Anxiety Inventory (STAI) is one of the most frequently used scales in anxiety research, although it is not a specific scale for dental anxiety. The inventory has 2 different scales, each with 20 items, showing the state and trait anxiety levels: STAI-state is used to determine a patient's current anxiety level, and STAI-trait is used to determine a patient's underlying (ongoing/personality) anxiety level. All 20 items are rated on a 4-point scale. The total score obtained can range from 20 to 80. STAI scores are commonly classified as "no or low anxiety" (20-37), "moderate anxiety" (38-44), and "high anxiety" (45-80). We used only STAI-S
Evaluation of anxiety with Dental Fear Survey(DFS) between groups preoperatively and postoperatively | 2 minutes
  DFS is a scale developed by Kleinknecht used to determine dental fear in different dimensions. This is a Likert-type scale with a score of 1-5. It has 20 items. It examines the level of fear in terms of dentist avoidance, somatic symptoms of fear, and fear of various applications in dentistry practice
Evaluation of anxiety with Modified Dental Anxiety Scale(MDAS) between groups preoperatively and postoperatively | 1 minute
  MDAS was developed by Humphris et al. by adding a question related to injection. The scale consists of five-point Likert-type rating with five options. The scoring in this scale varies between 5 and 25
Evaluation of anxiety with Visual Analog Scale (VAS) between groups preoperatively and postoperatively | 1 minute
  VAS is ideal for evaluating situations that cannot be measured using digital and oral information 25. In the present study, a scale comprising 100-mm closed-end line was used to measure the anxiety level. One end of the scale was labeled as "no anxiety" and the other end as "maximum anxiety imaginable."

CONTACTS AND LOCATIONS:
Overall Officials: Kevser Sancak, Study Chair — Ankara University Faculty of Dentısry
Locations (1):
- Ankara University dentisry of faculty, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Muglali M, Komerik N. Factors related to patients' anxiety before and after oral surgery. J Oral Maxillofac Surg. 2008 May;66(5):870-7. doi: 10.1016/j.joms.2007.06.662. PMID 18423273
- [Background] Jaakkola S, Rautava P, Alanen P, Aromaa M, Pienihakkinen K, Raiha H, Vahlberg T, Mattila ML, Sillanpaa M. Dental fear: one single clinical question for measurement. Open Dent J. 2009 Jul 28;3:161-6. doi: 10.2174/1874210600903010161. PMID 19672334
- [Background] Pell GJ. Impacted mandibular third molars: classification and modified techniques for removal. Dent Digest. 1933;39:330-338.
- [Background] Winter GB. Principles of exodontia as applied to the impacted mandibular third molar. American Medical Book Company; 1926.
- [Background] Ost L-g, Öst L-G, Skaret E. Cognitive behavioral therapy for dental phobia and anxiety. John Wiley & Sons; 2013